CLINICAL TRIAL: NCT04892758
Title: Replication of the P04334 Asthma Trial in Healthcare Claims Data
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Shirley Vichy Wang, Assistant Professor, Brigham and Women's Hospital
Other Study IDs: 2018P002966-DUP-P04334
Record Dates: First submitted 2021-05-14; First posted 2021-05-19 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Formoterol Fumarate; Mometasone Furoate; BID protein, human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Formoterol fumarate 10 mcg: Reference Group
  Interventions: Drug: Formoterol fumarate 10 mcg
- Mometasone furoate/formoterol fumarate combination MDI 200/10 mcg BID: Exposure Group
  Interventions: Drug: Mometasone furoate/formoterol fumarate combination MDI 200/10 mcg BID

INTERVENTIONS:
Drug: Formoterol fumarate 10 mcg — Formoterol fumarate 10 mcg dispensing claim is used as the reference group.
  Groups: Formoterol fumarate 10 mcg
Drug: Mometasone furoate/formoterol fumarate combination MDI 200/10 mcg BID — Mometasone furoate/formoterol fumarate combination MDI 200/10 mcg BID dispensing claim is used as the exposure group.
  Groups: Mometasone furoate/formoterol fumarate combination MDI 200/10 mcg BID

SUMMARY:
Investigators are building an empirical evidence base for real world data through large-scale replication of randomized controlled trials. The investigators' goal is to understand for what types of clinical questions real world data analyses can be conducted with confidence and how to implement such studies.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the RCT DUPLICATE initiative (www.rctduplicate.org) of the Brigham and Women's Hospital, Harvard Medical School. It is intended to replicate, as closely as is possible in healthcare insurance claims data, the trial listed below/above. Although many features of the trial cannot be directly replicated in healthcare claims, key design features, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial. Randomization is also not replicable in healthcare claims data but was proxied through a statistical balancing of measured covariates according to standard practice. Investigators assume that the RCT provides the reference standard treatment effect estimate and that failure to replicate RCT findings is indicative of the inadequacy of the healthcare claims data for replication for a range of possible reasons and does not provide information on the validity of the original RCT finding.

ELIGIBILITY:
Criteria:

Please see https://drive.google.com/drive/folders/1WD618wrywYjEaXzfLTcuK-VCcnb6b-gV for full code and algorithm definitions.

Eligible cohort entry dates:

Mometasone-furoate/formoterol was approved by FDA on June 24, 2010 for the management of asthma. The initial eligible cohort entry date was the first date after June 24, 2010 for both the databases investigated (IBM MarketScan, Optum CDM). The last date eligible as cohort entry date was the end of available data for IBM MarketScan and Optum

CDM. The following eligible cohort entry dates were included:

* Optum CDM: June 24, 2010 - June 30, 2020 (end of available data)
* IBM MarketScan: June 24, 2010- December 31, 2018 (end of available data)

Inclusion Criteria:

* ≥12 years of age
* A subject must have been using a medium daily dose of inhaled glucocorticosteroid (ICS) (either alone or in combination with a long-acting beta agonist (LABA)) for at least 12 weeks and must have been on a stable regimen (daily dose unchanged) for at least 2 weeks prior to Screening. Medium daily doses of ICS are defined as follows:

  1. >500 to 1000 mcg beclomethasone chlorofluorocarbon (CFC)
  2. >250 to 500 mcg beclomethasone hydrofluoroalkane (HFA)
  3. >600 to 1000 mcg budesonide dry powder inhaler (DPI)
  4. >1000 to 2000 mcg flunisolide
  5. >250 to 500 mcg fluticasone
  6. 400 mcg MF
  7. >1000 to 2000 mcg triamcinolone acetonide
* Diagnosis of asthma
* A female subject of childbearing potential must have been using a medically acceptable, adequate form of birth control.

Exclusion Criteria:

* A subject who experiences an occurrence of any clinical deterioration of asthma that results in emergency treatment, hospitalization due to asthma, or treatment with additional, excluded asthma medication (other than SABA) as judged by the clinical investigator at any time from the Screening Visit up to and including the Baseline Visit
* Emergency room treatment for asthma deterioration requiring systemic corticosteroid therapy or hospitalization for management of airway obstruction within the 3 months before baseline
* A subject who is a smoker or ex-smoker and has smoked within the previous year or has had a cumulative smoking history >10 pack-years
* Visible evidence of oropharyngeal candidiasis at baseline or earlier

Ages: 12 Years to 120 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This study will involve a new user, parallel group, propensity score-matched, retrospective cohort design comparing mometasonefuroate/formoterol 200/10ug with formoterol 12 ug in patients with persistent asthma previously receiving medium-dose inhaled corticosteroids. The patients will be required to have continuous enrollment during a baseline period of 180 days before initiation of mometasone-furoate/formoterol or formoterol. (Note: the formoterol dose used in the trial was 10ug ; in the replication, we will use the market available dose which is 12 ug).
Sampling Method: Non-Probability Sample
Enrollment: 10288 (Actual)
Dates: Start 2020-10-29 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

PRIMARY OUTCOMES:
Time to first asthma exacerbation | Through study completion (a median of 134-147 days)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Wang, PhD, ScM, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT04892758/Prot_SAP_001.pdf